CLINICAL TRIAL: NCT06304389
Title: Effect of Blue Light on Vagus Nerve Stimulation in Patients With Refractory Epilepsy
Acronym: BLUELIGHTVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BLUELIGHT-VNS
Record Dates: First submitted 2023-04-18; First posted 2024-03-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Evoked Potentials

STUDY DESIGN:
Intervention Model Description: Patients with refractory epilepsy (divided in non responders & responders), and healthy subjects
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with refractory epilepsy (Experimental): Patients will not receive any drugs, but will participate to experiments involving electroencephalograpy, pupillometry and light administration.
  Interventions: Other: electroencephalography, electrocardiogram, pupillometry, evoked potentials, light administration
- Healthy subjects (Experimental): Subjects will not receive any drugs, but will participate to experiments involving electroencephalograpy, pupillometry and light administration.
  Interventions: Other: transcutaneous vagus nerve stimulation, electroencephalography, pupillometry, electrocardiogram, light administration

INTERVENTIONS:
Other: electroencephalography, electrocardiogram, pupillometry, evoked potentials, light administration — Recording of the electrical activity of the brain, of the heart. Pupil size will be analyzed. The effect of blue light administration will be assessed on those parameters.
  Arms: Patients with refractory epilepsy
Other: transcutaneous vagus nerve stimulation, electroencephalography, pupillometry, electrocardiogram, light administration — Transcutaneous vagus nerve stimulation will be performed in helathy subjects, as well as the recording of the electrical activity of the brain, and of the heart. Pupil size will be analyzed. The effect of blue light administration will be assessed on those parameters.
  Arms: Healthy subjects

SUMMARY:
Vagus nerve stimulation (VNS) is an adjunctive treatment for refractory epilepsy. Although widely used, there is still a substantial number of patients with insufficient response. Light, and particularly blue light, can stimulate alertness, attention and cognition through modulation of anatomical targets which are common to the vagal afferent network. This project aims at understanding how exposure to blue enriched light may influence VNS effects in patients with refractory epilepsy by exploring the modulation of a series of biomarkers of VNS action. This could possibly lead to new therapeutic strategies to increase efficacy of VNS.

ELIGIBILITY:
Inclusion Criteria:

Patients:

VNS implanted since at least 3 months age >18-60 years; IQ >55 on Wechsler scale (normal status or mild cognitive impairment)

healthy participants aged between 18 and 35 years without any medical history (neurological / psychiatric disease)

Exclusion criteria:

Patients:

other medical implanted devices than VNS, ocular diseases

Helthy participants:

medical implanted devices, cerebral trauma, ocular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Effect of blue light on VNS biomarkers | 4 years
  Blue light increases VNS induced electroencephalogram desynchronisation in implanted patients
Effect of blue light on VNS biomarkers | 4 years
  Blue light increases P300 amplitude in VNS implanted patients
Effect of blue light on VNS biomarkers | 4 years
  Blue light increases VNS (or tVNS) induced pupil dilation (in patients & healthy subjects).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Woluwe-Saint-Lambert, Belgium